CLINICAL TRIAL: NCT03508921
Title: Comparison of Methods for Prevention of Urinary Tract Infection Following Botox Injection: a Non-Inferiority Trial
Brief Title: Comparison of Methods for Prevention of Urinary Tract Infection Following Botox Injection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination due to recruitment and follow-up challenges during the pandemic
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Allergan Foundation (Other); Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (Other)
Responsible Party: Principal Investigator, Melissa Kaufman, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00011112222
Record Dates: First submitted 2018-03-13; First posted 2018-04-26 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Overactive Bladder; Urinary Tract Infections
Keywords: Onabotulinumtoxin
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periprocedural Antibiotics Only (Experimental): Patients receive a one-time dose of antibiotics at the time of injection, prior to injection.
  Interventions: Drug: Periprocedural Antibiotics; Procedure: Injection of OnabotulinumtoxinA (BTX-A)
- Extended Antibiotics (Experimental): Patients receive a peri-procedural dose of antibiotics and an extended (3-day) course of antibiotics to be taken post-procedurally.
  Interventions: Drug: Periprocedural Antibiotics; Drug: Extended Antibiotics; Procedure: Injection of OnabotulinumtoxinA (BTX-A)

INTERVENTIONS:
Drug: Periprocedural Antibiotics — One the day of injection, after eligibility is determined and consent obtained, research staff will refer to the randomization list to determine to which arm the patient is randomized. Patients randomized to the "Procedural Antibiotics Only" arm will receive a single dose of trimethoprim/sulfamethoxazole (800/160mg) peri-procedurally at the time of the first injection.
  Other Names: trimethoprim/sulfamethoxazole
Drug: Extended Antibiotics — Patients randomized to the "Extended Antibiotics" arm will receive one dose of trimethoprim/sulfamethoxazole peri-procedurally and additionally be prescribed trimethoprim/sulfamethoxazole twice daily for three days. Patients who are allergic will receive amoxicillin/clavulanic acid (875/125mg) twice daily for three days. If allergic to both of the above antibiotics, patients will receive 100mg nitrofurantoin BID for three days.
  For their second injection, they will receive peri-procedural antibiotics only.
  Other Names: trimethoprim/sulfamethoxazole
  Arms: Extended Antibiotics
Procedure: Injection of OnabotulinumtoxinA (BTX-A) — Patients will receive injection of OnabotulinumtoxinA (BTX-A) per standard clinic practice protocol. All patients will undergo injection per a standardized protocol of 1ml injection per site at a concentration of 10 units/ml.

SUMMARY:
Injection of OnabotulinumtoxinA (BTX-A) into the bladder is a widely used treatment option for patients with overactive bladder who have failed medical therapy. Urinary tract infection is the most common side effect of this procedure and therefore antibiotics are given around the time of injection in order to prevent these events. While antibiotics are commonly given at the time of injection, the duration of these antibiotic regimens are variable. The investigators propose a study to investigate different antibiotic protocols and their affect on the rate of urinary tract infection after injection.

DETAILED DESCRIPTION:
Intravesical injection of OnabotulinumtoxinA (BTX-A) is a widely practiced third line therapy for non-neurogenic overactive bladder (OAB). However, a paucity of data exists regarding urinary tract infections (UTI), the most common adverse event following injection. The investigators propose a randomized, controlled cross-over trial to investigate the utility of commonly practiced antibiotic protocols and simultaneously derive information regarding risk factors for post-procedural UTIs and their affect on treatment efficacy.

The investigators plan to initiate a prospective, randomized non-inferiority cross-over trial, in which a participant receives peri-procedural antibiotics exclusively at the time of one injection, and then at a subsequent injection, completes a three-day course of antibiotics post-operatively in addition to the peri-procedural dose. Enrollment is planned to achieve a total of 68 participants. Participants will be evaluated at 3 weeks and 3 months following injection to identify adverse events and treatment success. Inter-injection time will be measured and used a surrogate for efficacy over multiple injections.

These results, in addition to filling a void in current literature regarding the increasingly utilized treatment with BTX-A, have the potential to modify clinical practice regarding antibiotic use and decrease rates of adverse events. The means to stratify patients based on their specific risk of UTI may be used to facilitate antibiotic stewardship and improve patient outcomes.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years of age
* Medication refractory OAB, identified per American Urological Association guidelines

Exclusion criteria:

* Post void residual urine >150ml on two occasions
* Untreated, symptomatic UTI
* Comorbid neurological conditions, including spinal cord injury, systemic neurologic illnesses (i.e. multiple sclerosis, Parkinson's disease) or central nervous system disease (i.e. brain tumor, stroke)
* Prior pelvic irradiation
* Current or prior bladder malignancy
* Hematuria lacking a clinically appropriate evaluation
* Chronic indwelling or intermittent catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kaufman, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment halted
Pre-assignment Details: 22 participants were randomized. Data is reported only for the 17 participants who fully completed both injections and all follow-up visits.
Groups:
- Periprocedural Antibiotics Only, Then Extended Antibiotics: All patients will undergo an intravesical injection of OnabotulinumtoxinA (Botox ®, BTX-A) per a standardized protocol of 1ml injection per site at a concentration of 10 units/ml at Visit 1 and a second injection at Visit 2.
  Participants will also receive:
  * Periprocedural Antibiotics Only: At Visit 1, patients will receive a single dose of trimethoprim/sulfamethoxazole (800/160mg) peri-procedurally
  * Extended antibiotics: At Visit 2, patients will receive one dose of trimethoprim/sulfamethoxazole periprocedurally and additionally be prescribed trimethoprim/sulfamethoxazole twice daily for three days. Patients who are allergic will receive amoxicillin/clavulanic acid (875/125mg) twice daily for three days. If allergic to both of the above antibiotics, patients will receive 100mg nitrofurantoin BID for three days
- Extended Antibiotics, Then Periprocedural Antibiotics Only: All patients will undergo an intravesical injection of OnabotulinumtoxinA (Botox ®, BTX-A) per a standardized protocol of 1ml injection per site at a concentration of 10 units/ml at Visit 1 and a second injection at Visit 2.
  Participants will also receive:
  * Extended antibiotics: At Visit 1, patients will receive one dose of trimethoprim/sulfamethoxazole periprocedurally and additionally be prescribed trimethoprim/sulfamethoxazole twice daily for three days. Patients who are allergic will receive amoxicillin/clavulanic acid (875/125mg) twice daily for three days. If allergic to both of the above antibiotics, patients will receive 100mg nitrofurantoin BID for three days
  * Periprocedural Antibiotics Only: At Visit 2, patients will receive a single dose of trimethoprim/sulfamethoxazole (800/160mg) peri-procedurally
Period: Overall Study
Arm/Group | Periprocedural Antibiotics Only, Then Extended Antibiotics | Extended Antibiotics, Then Periprocedural Antibiotics Only
Started | 10 | 12
Completed | 6 | 11
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Population: 22 participants were randomized. Data is reported only for the 17 participants who fully completed both injections and all follow-up visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | Periprocedural Antibiotics Only, Then Extended Antibiotics | Extended Antibiotics, Then Periprocedural Antibiotics Only | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Post Procedural- Urinary Tract Infection
Description: Number of participants with post procedural- urinary tract infection 3 weeks after injections, measured by a urine culture and defined as a urine culture with >10^5 bacterial colonies in the setting of urinary symptoms.
Time Frame: 3 weeks post-injection
Population: Data is reported only for the 17 participants who fully completed both injections and all follow-up visits.
Measure: Number; unit: participants
Arm/Group | Periprocedural Antibiotics Only, Then Extended Antibiotics | Extended Antibiotics, Then Periprocedural Antibiotics Only
Number analyzed (Participants) | 6 | 11
participants
  Visit 1: 3 weeks post-injection | 0 | 1
  Visit 2: 3 weeks post-injection | 0 | 2

2. Secondary Outcome: Urinary Retention
Description: Number of participants with urinary retention > 250 cc post-procedurally as measured by post void residual volume using a bladder scanner in clinic.
Time Frame: 3 weeks post-injection
Population: Data is reported only for the 17 participants who fully completed both injections and all follow-up visits.
Measure: Number; unit: participants
Arm/Group | Periprocedural Antibiotics Only, Then Extended Antibiotics | Extended Antibiotics, Then Periprocedural Antibiotics Only
Number analyzed (Participants) | 6 | 11
participants
  Visit 1: 3 weeks post-injection | 1 | 3
  Visit 2: 3 weeks post-injection | 0 | 3

3. Secondary Outcome: Recurrent Urinary Tract Infection
Description: Number of participants with 3 or greater post procedural- urinary tract infection after injections, measured by a urine culture and defined as a urine culture with >10^5 bacterial colonies in the setting of urinary symptoms.
Time Frame: 3 weeks post injection
Population: Data is reported only for the 17 participants who fully completed both injections and all follow-up visits.
Measure: Number; unit: participants
Arm/Group | Periprocedural Antibiotics Only, Then Extended Antibiotics | Extended Antibiotics, Then Periprocedural Antibiotics Only
Number analyzed (Participants) | 6 | 11
participants
  Visit 1: 3 weeks post-injection | 0 | 0
  Visit 2: 3 weeks post-injection | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months following second injection, 6 month total time frame from randomization
Description: Data is reported only for the 17 participants who fully completed both injections and all follow-up visits.
Groups:
- Periprocedural Antibiotics Only: Patients who received a single dose of trimethoprim/sulfamethoxazole (800/160mg) peri-procedurally.
- Extended Antibiotics: Patients who received one dose of trimethoprim/sulfamethoxazole periprocedurally and additionally were prescribed trimethoprim/sulfamethoxazole twice daily for three days. Patients who are allergic received amoxicillin/clavulanic acid (875/125mg) twice daily for three days. If allergic to both of the above antibiotics, patients received 100mg nitrofurantoin BID for three days.
Arm/Group | Periprocedural Antibiotics Only | Extended Antibiotics
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Early termination due to recruitment and follow-up challenges during the pandemic resulting in failure to accrue statistically significant sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03508921/Prot_SAP_003.pdf